CLINICAL TRIAL: NCT01015040
Title: A Phase 1, Open-Label, Randomized, Single Dose, 3-Way Crossover Study to Address the Relative Bioavailability of Solifenacin Liquid Suspension 10mg (Fed and Fasting) Versus the VESIcare (Solifenacin Succinate) 10 mg Tablet (Fasting) in Healthy Volunteers
Brief Title: Relative Bioavailability Study of Solifenacin Succinate Liquid Suspension (Fed and Fasting) Versus VESIcare Tablet (Fasting) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sr. Manager Clinical Trials Registry, Astellas Pharma Global Development
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 905-CL-066
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Bioavailability of Solifenacin Succinate; Pharmacokinetics of Solifenacin Succinate; Healthy Volunteers
Keywords: solifenacin succinate; VESIcare; Healthy Volunteers
MeSH Terms: interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- solifenacin succinate tablet (fasting) (Active Comparator)
  Interventions: Drug: solifenacin succinate tablet
- solifenacin succinate suspension (fasting) (Experimental)
  Interventions: Drug: solifenacin succinate suspension
- solifenacin succinate suspension (fed) (Experimental)
  Interventions: Drug: solifenacin succinate suspension

INTERVENTIONS:
Drug: solifenacin succinate suspension — Oral
  Other Names: YM905
  Arms: solifenacin succinate suspension (fasting); solifenacin succinate suspension (fed)
Drug: solifenacin succinate tablet — Oral
  Other Names: VESIcare; YM905
  Arms: solifenacin succinate tablet (fasting)

SUMMARY:
The objective of the study is to compare the relative bioavailability and pharmacokinetics of solifenacin succinate suspension versus tablet.

DETAILED DESCRIPTION:
All subjects will participate in each treatment separated by a minimum (=> minimum) of 13 days between dosing.

In the two fasting periods, each subject will receive solifenacin succinate orally in each treatment period following a minimum 10 hour fast from food and beverages. In the fed condition, each subject will receive the suspension within 30 minutes of the start of breakfast.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject weighing at least 45 kg with a Body Mass Index (BMI) of 18-32 kg/m2, inclusive
* If female, subject is at least 2 years postmenopausal, surgically sterile or practicing effective birth control and is not lactating or pregnant
* Medically healthy, with a normal 12-lead electrocardiogram (ECG)
* Good venous access in both arms

Exclusion Criteria:

* History of any clinically significant disease or malignancy excluding non-melanoma skin cancer
* Known hypersensitivity to VESIcare® or any of the excipients in the formulations, or a history of severe allergic or anaphylactic reactions
* History of alcoholism or substance abuse within past 2 years
* Has used tobacco-containing products and nicotine or nicotine containing products within six months
* Supine mean systolic blood pressure < 90 or > 160 mmHg and a mean diastolic blood pressure < 50 or > 90 mmHg, or pulse rate < 40 or > 100 beats per minute
* Positive test for hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg)
* Known positive for human immunodeficiency virus (HIV) antibody
* Clinical laboratory tests outside the normal limits
* Treatment with prescription or non-prescription drugs, including complementary and alternative medicines or over-the-counter medications, with the exception of oral contraceptives, hormone replacement therapy, and occasional use of acetaminophen within 14 days prior to Day 1
* Inability to abstain from alcohol or caffeine use for 48 hours prior to the administration of the first dose of study drug and throughout the duration of the study or from grapefruit, Seville oranges, star fruit, or any products containing these items from 72 hours prior to the administration of the first dose of study drug and throughout the duration of the study
* Donated one unit of blood or more, has had significant blood loss, or received a transfusion of any blood or blood products within 60 days or has donated plasma within 7 days prior to study check-in
* Any clinically significant history of gastrointestinal symptoms such as nausea, abdominal discomfort or upset, or heartburn in the four weeks prior to study check-in or a history of any gastrointestinal surgery except for appendectomy or cholecystectomy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Serum solifenacin succinate pharmacokinetics (PK) parameters | Periods 1, 2 and 3 Days 1-11

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- West Bend, Wisconsin, United States